CLINICAL TRIAL: NCT06322602
Title: Ommaya Reservoir Placement at the Time of Biopsy for Longitudinal Biomarker Collection
Brief Title: Ommaya Reservoir Placement at the Time of Biopsy for Longitudinal Biomarker Collection in Patients With Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-009112; NCI-2024-01762 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); R33NS122096 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms | interventions — Spinal Puncture; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ommaya reservoir placement (Experimental): Patients undergo Ommaya reservoir placement during standard of care biopsy. Patients then undergo extraction of CSF while on study. Patients may also optionally undergo lumbar puncture while on study. Patients also undergo CT or MRI on study.
  Interventions: Procedure: Intracranial Catheter Placement; Procedure: Lumbar Puncture; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Intracranial Catheter Placement — Undergo Ommaya reservoir placement
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; spinal tap
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Cerebrospinal Fluid Collection; CSF Collection; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; Structural MRI; sMRI

SUMMARY:
This observational trial evaluates the use of Ommaya reservoir placed during a biopsy to collect biomarkers longitudinally in patients with brain tumor. A biomarker is a measurable indicator of the severity or presence of the disease state. An Ommaya reservoir is a small device that's implanted under the scalp. It allows the doctor to take samples of cerebrospinal fluid (CSF) in the future without doing a spinal tap. The identification of biomarkers in CSF is rapidly emerging as a promising minimally invasive approach for monitoring tumor growth and response to therapy. In the future, these biomarkers may be used to help determine what treatments could be most effective and how well a tumor has responded to prior therapy. Currently, limited long-term access to CSF has made it difficult for studies to learn if collecting CSF at different points in the treatment process is useful. Having an Ommaya reservoir placed during a biopsy may allow for longitudinal biomarker collection in patients with brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiographic evidence suggesting a diagnosis of a brain tumor
* Planned biopsy for suspected or previously diagnosed brain tumor as part of routine clinical care at Mayo Clinic (Rochester, Minnesota [MN])
* Willingness of the patient to provide informed consent
* Patient is willing to have their Ommaya sampled on at least 2 future occasions
* Patients is willing to have CSF banked through the neuro-oncology biorepository (requires a separate signature)

Exclusion Criteria:

* Adults lacking capacity to consent
* Vulnerable populations including pregnant women, prisoners, and individuals < 18 years old
* Patients who are not appropriate candidates for biopsy due to current or past medical history or uncontrolled current illness
* Prior history of any wound infection
* Any patient who the surgeon feels is not an optimal candidate for Ommaya reservoir placement. Such reasons may include, but will not be limited to, surgical anatomy, clinical evidence of immunosuppression, and/or elevated risk of wound infection due to diabetes, smoking history, morbid obesity, or any other concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Ommaya reservoir placement | Up to 5 years
  Will be assessed based on the percent of patients for whom an Ommaya reservoir is successfully placed at the time of tissue biopsy without attributable complication.

SECONDARY OUTCOMES:
Utility of Ommaya reservoir | Up to 5 years
  Will be assessed based on the percent of patients for whom multiple (2 or more) cerebrospinal fluid (CSF) samples are successfully obtained as a result of their participation in this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Terry C. Burns, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials